CLINICAL TRIAL: NCT01176799
Title: Phase II Randomized Study of Doxorubicin and Cyclophosphamide With or Without Intermittent Sunitinib in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer Patients With Measurable Primary Breast Tumor
Brief Title: Randomized Study of Doxorubicin and Cyclophosphamide With or Without Intermittent Sunitinib in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer Patients With Measurable Primary Breast Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR01/09/10
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer patients with measurable primary breast cancer tumor.
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Control Arm (Active Comparator): Doxorubicin - 60mg/m2 day 1
  Cyclophosphamide
  -600mg/m2 day1, every 3 weeks x 4 cycles
  Interventions: Drug: Arm A
- Arm B: Experimental (Experimental): Days -13 (or -7) to day 0 (total 7 or 14 days) - oral sunitinib daily Cycle 1: day 1 - Cycle 1 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 2: day 1 - Cycle 2 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 3: day 1 - Cycle 3 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 4: day 1 - Cycle 4 AC (60/600mg/m2)
  Interventions: Drug: Arm B

INTERVENTIONS:
Drug: Arm A — Doxorubicin 60mg/m2 day 1 Cyclophosphamide 600mg/m2 day1, every 3 weeks x 4 cycles
  Other Names: Control Arm; Doxorubicin and Cyclophosphamide
  Arms: Arm A: Control Arm
Drug: Arm B — Days -13 (or -7) to day 0 (total 7 or 14 days) - oral sunitinib daily Cycle 1: day 1 - Cycle 1 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 2: day 1 - Cycle 2 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 3: day 1 - Cycle 3 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 4: day 1 - Cycle 4 AC (60/600mg/m2)
  Other Names: Experimental Arm:; Sunitinib and doxorubicin and cyclophosphamide (AC)
  Arms: Arm B: Experimental

SUMMARY:
This is a single-centre, phase II randomized study of doxorubicin and cyclophosphamide (AC) with or without intermittent sunitinib in patients with measurable primary breast cancer who are receiving pre-operative chemotherapy.

A lead-in phase I study was built into this protocol to determine the dose and duration of sunitinib that may achieve the desired effects of normalizing tumor vasculature prior to chemotherapy administration.

A total of 64 patients with measurable primary tumor will be enrolled for the Phase II part of the study. Eligible patients will be randomized 1:1 to either arm A or arm B. Patients will be stratified according to metastatic status (metastatic vs non-metastatic) and presence or absence of clinical T4 disease.

Arm A (Control arm):

Doxorubicin 60mg/m2 day 1 Cyclophosphamide 600mg/m2 day1, every 3 weeks x 4 cycles

Arm B (Experimental arm):

Days -13 (or -7) to day 0 (total 7 or 14 days) - oral sunitinib daily (duration and dose as determined from the lead-in phase I study) Cycle 1: day 1 - Cycle 1 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 2: day 1 - Cycle 2 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 3: day 1 - Cycle 3 AC (60/600mg/m2); days 15-21 - oral sunitinib daily Cycle 4: day 1 - Cycle 4 AC (60/600mg/m2)

DCE-MRI scan will be performed serially to determine tumor response and change in tumor vascular parameters for each enrolled subject:

Patient will be evaluated weekly for toxicity assessments and full blood count during cycle 1, and on days 1 and 15 of each subsequent cycle. In addition, patients in Arm B will be evaluated weekly during the first two weeks of sunitinib administration prior to cycle 1 AC.

DETAILED DESCRIPTION:
Special tests Blood sampling

* Germline DNA at baseline for pharmacogenetics analysis.
* Pharmacokinetic sampling for doxorubicin and cyclophosphamide on day 1, cycle 1 of AC administration.
* Pharmacokinetic sampling for sunitinib at baseline and weekly during the first course of sunitinib for subjects in Arm B before the sunitinib dose on that day.
* Serial plasma samples for proteomics analysis and for analysis of soluble angiogenic factors
* Serial whole blood for gene expression analysis
* Serial blood samples for circulating tumor and circulating endothelial cells
* DNA will be extracted from collected snap-frozen and/or paraffin-embedded tumor tissue sections (pre- and post-treatment) and plasma (pre- and post-treatment taken for plasma biomarker analysis). Primary tumor and circulating tumor DNA will be genotyped for cancer genes of interest that may influence cancer prognosis and/or treatment response.

Tumor core biopsy Arm A: Performed at baseline, approximately 3 weekly after cycle 1 AC but before cycle 2 AC, and upon completion of 4 cycles of AC, for a total of 3 tumor core biopsies Arm B: Performed at baseline, after completing the first course of sunitinib and before cycle 1 AC, approximately 3 weekly after cycle 1 AC but before cycle 2 AC, and upon completion of 4 cycles of AC, for a total of 4 tumor core biopsies.

The final biopsy may be obtained at surgery if the patient is scheduled for lumpectomy or mastectomy. The tumor cores will be stored in liquid nitrogen for subsequent DNA, RNA and protein extraction for biomarker studies including gene expression and proteomics analyses. Three to four samples will be obtained at each time point, and one tumor core at each time point will be stored in formalin and paraffin-embedded for immunohistochemistry analysis of biomarkers.

Note: Tumor biopsies, imaging and blood collection that are to be conducted after completing the first course of sunitinib may be carried out as early as 2 days before the last dose of sunitinib in the first course for logistics reasons.

ELIGIBILITY:
Inclusion Criteria:

* Female, age >= 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* T2-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper.
* Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  * Bone marrow:
* Absolute neutrophil (segmented and bands) count (ANC) >=1.5 x 109/L
* Platelets >= 100 x 109/L

  * Hepatic:
* Bilirubin <= 1.5 x upper limit of normal (ULN),
* ALT or AST <= 2.5x ULN, (or <= 5 X with liver metastases)

  * Renal:
* Creatinine <= 1.5x ULN
* Left ventricular ejection fraction >=50%
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (e.g., intrauterine device, birth control pills, or barrier device) during and for three months after the study.Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Prior treatment for locally advanced or metastatic breast cancer.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Known history of systemic connective tissue diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis), vasculitides (e.g., giant cell arteritis, Kawasaki disease, Wegener's granulomatosis, Churg-Strauss disease) or sickle cell disease.
* Known history of renal impairment, defined as a Glomerular Filtration Rate (GFR) of less than 30ml/minute.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | 12 weeks
  To compare the pathological complete response rate of doxorubicin/cyclophosphamide with or without intermittent sunitinib in the first-line pre-operative setting in breast cancer in the Phase II part of the study.

SECONDARY OUTCOMES:
clinical response rate | 12 weeks
  To compare the clinical response rate (complete and partial response) and progression-free survival in patients treated with 4 cycles of doxorubicin/cyclophosphamide with or without intermittent sunitinib in the first-line pre-operative setting in breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore